CLINICAL TRIAL: NCT06838494
Title: Utilization of Immersive Virtual Reality in Cognitive Stimulation Therapy (IVR-CST) for Elderly with Mild Cognitive Impairment: a Randomized Controlled Pilot Study
Brief Title: Using Immersive Virtual Reality for Cognitive Therapy in Elderly with Mild Cognitive Impairment
Acronym: VR-CST-MCI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The University of Hong Kong (Other); University of Reading (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20241010009; 22231471 (Other Grant/Funding Number: Health and Medical Research Fund)
Record Dates: First submitted 2025-02-07; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: Mild Cognitive Impairment (MCI); Cognitive stimulation therapy; immersive reality; Eye-tracking
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IVR-CST Group (Experimental)
  Interventions: Behavioral: IVR-CST (Immersive Virtual Reality Cognitive Stimulation Therapy)
- Conventional CST Group (Active Comparator)
  Interventions: Behavioral: Intervention Name: Conventional CST (Cognitive Stimulation Therapy)

INTERVENTIONS:
Behavioral: IVR-CST (Immersive Virtual Reality Cognitive Stimulation Therapy) — IVR-CST involves 14 sessions of cognitive stimulation therapy conducted twice a week in a virtual reality environment. Each session lasts approximately 45 minutes and utilizes head-mounted displays (HMDs) to immerse participants in engaging, themed activities. The therapy aims to enhance cognitive function and social interaction through interactive and stimulating virtual experiences tailored for individuals with mild cognitive impairment (MCI).
  Arms: IVR-CST Group
Behavioral: Intervention Name: Conventional CST (Cognitive Stimulation Therapy) — Conventional CST consists of 14 sessions of cognitive stimulation therapy conducted twice a week, each lasting about 45 minutes. In this arm, participants engage in group activities using physical materials, such as photos, pictures, and real objects, rather than virtual reality. The therapy focuses on providing cognitive stimulation through discussions and activities designed to improve cognitive function and social engagement among individuals with mild cognitive impairment (MCI).
  Arms: Conventional CST Group

SUMMARY:
The proposed study aims to investigate the potential of IVR-CST in improving cognition of people with MCI, and as well the association of eye movement during therapy and treatment outcomes of IVR-CST. Four research questions have been proposed and listed as follows:

1. Is IVR-CST a feasible treatment for elderly with MCI?
2. Is IVR-CST an efficacious treatment for improving cognition of elderly with MCI?
3. Is IVR-CST more efficacious than conventional CST (i.e., without IVR) in improving the cognition of elderly with MCI?
4. Is eye-tracking data collected during therapy associated with treatment outcomes of IVR CST?

ELIGIBILITY:
Inclusion Criteria:

1. elderly aged 60 years or above,
2. a diagnosis of MCI made by a psychiatrist, or a score of 16-21 out of 30 in the Hong Kong Brief Cognitive Test (HKBC, 31), with upper and lower cutoff scores for MCI as suggested by the test. HKBC has been validated in Hong Kong with satisfactory sensitivity (0.88) and specificity ((0.81) in differentiating subjects with MCI and healthy individuals,
3. ability to speak and comprehend Cantonese,
4. normal or corrected-to-normal binocular vision and hearing,
5. absence of physical illness/disability to prevent them from IVR-CST participation, 6, compatible with IVR exposure in the 10-minute IVR trial without major signs of cybersickness, based on the symptoms given in the Simulator Sickness Questionnaire

Exclusion Criteria:

1. concurrent participation in other clinical therapy trials,
2. incompatibility with IVR exposure such as complaints of nausea, headache, or other severe discomforts during trial use,
3. a diagnosis of dementia or other psychiatric/neurological diseases such as depression, stroke, brain trauma, Parkinson's disease
4. hearing/visual/upper limb impairments that hinder CST/IVR-CST participation,
5. prior CST treatment,
6. Use of medication for MCI/dementia, e.g., aducanumab

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-07-03 (Estimated); Primary Completion 2026-10-02 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Hong Kong Montreal Cognitive Assessment (HK-MoCA) | From 1-week pre-intervention to 13 weeks post-intervention
  Hong Kong Montreal Cognitive Assessment (HK-MoCA) Measurement of global cognition in participants, covering various cognitive domains such as visuo-spatial skills, executive functions, attention, memory, language, and orientation. The total score ranges from 1-30, with higher score indicating better performance.
Digit Span Forward and Backward Tasks | From 1-week pre-intervention to 13 weeks post-intervention
  Assessment of working memory capacity, predicting progression from MCI to dementia. The test will start from 1 digit with increasing number of digit to increase level of difficulty.
Verbal Fluency of Semantic Category | From 1-week pre-intervention to 13 weeks post-intervention
  Evaluation of semantic integrity, cognitive flexibility, and executive function by measuring the number of items correctly produced in one minute across different semantic categories (animals, fruits, transportation).

SECONDARY OUTCOMES:
Chinese Version of the Modified Barthel Index | From 1-week pre-intervention to 13 weeks post-intervention
  Assessment of the level of independence in activities of daily living, including grooming, feeding, mobility, toileting, and more. The test score ranges from 1-100 with higher scores indicating better performance.
Hong Kong Lawton Instrumental Activities of Daily Living Scale | From 1-week pre-intervention to 13 weeks post-intervention
  Evaluation of independence in performing community-living skills, such as cooking, household management, and shopping. The test score ranged from 0-18 and a higher score indicates better performance.
Feasibility Outcomes and Users' Experience | Throughout the intervention period (from weeks 1-7 of intervention)
  Objective measures of feasibility, including the number of adverse events and technical issues during the intervention, as well as adherence to the intervention protocol (actual duration and number of sessions conducted vs. scheduled).
Semi-Structured Interview for IVR-CST Group | Immediately post-intervention
  Post-therapy interview assessing comfort levels, presence of adverse effects (e.g., cybersickness), and the impact of therapy on daily functions. Conducted by a trained research assistant in a quiet clinical room, with the session audio-taped.

CONTACTS AND LOCATIONS:
Overall Officials: Winsy WS Wong, PHD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The IPD, together with the study protocol, will be shared in an open-access data repository (e.g., OSF).
Supporting Information: Study Protocol, ICF
Time Frame: Data will be shared starting from three months after manuscript publication.
Access Criteria: The IPD and study protocol will be shared in an open-access data repository without restrictions.

REFERENCES:
- [Derived] Wong WWS, Wong GHY, Choy JCP, Pui Li DS, Lo YL. Utilization of Immersive Virtual Reality in Cognitive Stimulation Therapy (IVR-CST) for elderly with mild cognitive impairment: A randomized controlled pilot study protocol. PLoS One. 2025 Aug 26;20(8):e0330686. doi: 10.1371/journal.pone.0330686. eCollection 2025. PMID 40857307